CLINICAL TRIAL: NCT00118924
Title: Phase 1 Study of the Safety and Immunogenicity of Tick-Borne Langat/Dengue 4 Chimera (LGT(TP21)/DEN4), a Live Attenuated Vaccine for Tick-Borne Encephalitis
Brief Title: Safety of and Immune Response to a Tick-Borne Encephalitis Vaccine (LGT(TP21)/DEN4) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Anna Durbin, MD, Center for Immunization Research, Johns Hopkins School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 182; H.22.03.09.26.B2
Record Dates: First submitted 2005-07-08; First posted 2005-07-12 (Estimated); Last update posted 2008-01-21 (Estimated); Status verified 2008-01

CONDITIONS: Tick-Borne Encephalitis
Keywords: Dengue Vaccine; Tick-Borne Illnesses; Flavivirus
MeSH Terms: conditions — Encephalitis, Tick-Borne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): One subcutaneous vaccination with a 10^3 PFU dose of LGT(TP21)/DEN4 vaccine given in the deltoid region of either arm. A second booster vaccination will be given 6 months after the first vaccination.
  Interventions: Biological: LGT(TP21)/DEN4
- 2 (Experimental): One subcutaneous vaccination with a 10^5 PFU dose of LGT(TP21)/DEN4 vaccine given in the deltoid region of either arm. A second booster vaccination will be given 6 months after the first vaccination. This arm may enroll after Arm 1 depending on the immunological response of Arm 1.
  Interventions: Biological: LGT(TP21)/DEN4
- 3 (Placebo Comparator): One subcutaneous vaccination with a placebo vaccine given in the deltoid region of either arm. A second placebo vaccination will be given 6 months after the first vaccination.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: LGT(TP21)/DEN4 — Live attenuated LGT(TP21)/DEN4 vaccine (one of two doses)
  Arms: 1; 2
Biological: Placebo — Placebo for LGT(TP21)/DEN4 vaccine
  Arms: 3

SUMMARY:
Tick-borne encephalitis (TBE) is a viral illness common in the Northern Hemisphere, especially Europe and Asia. TBE infection may lead to central nervous system problems and death. The purpose of this study is to test the safety of and immune response to a TBE vaccine in healthy adults. The vaccine is related to a live attenuated virus developed against dengue virus infection.

DETAILED DESCRIPTION:
TBE is a common illness in Europe and Asia, where it is usually associated with mild illness but sometimes leads to long-term symptoms and even death. This study will evaluate the safety and immunogenicity of a live attenuated chimeric virus, LGT(TP21)/DEN4, which is derived from the Langat flavivirus and DEN4 dengue virus serotypes.

Each volunteer will be involved in the study for 180 days. Participants in Cohort 1 will be randomly assigned to receive LGT(TP21)/DEN4 or placebo at study entry. Cohort 2 will begin only after safety review of all participants in Cohort 1. Participants in Cohort 2 will receive a higher dose of LGT(TP21)/DEN4 or placebo.

After vaccination, participants will be asked to monitor their temperatures every day for 16 days and on Day 19. Study visits will occur every other day after vaccination until Day 16, followed by 5 additional visits at selected days through Day 180. Blood collection and a targeted physical exam will occur at each study visit. Some participants will be asked to undergo a skin biopsy or additional blood collection at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* Willing and available to be followed for the duration of the study
* Willing to use acceptable means of contraception
* Good general health

Exclusion Criteria:

* Pregnancy or breastfeeding
* Clinically significant neurologic, heart, lung, liver, rheumatologic, autoimmune, or kidney disease
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the ability of the volunteer to understand and cooperate with the study
* Blood disease
* History of migraine headaches
* History of encephalitis
* Alcohol or drug use that has caused medical, occupational, or family problems within 12 months prior to study entry
* History of severe allergic reaction or anaphylaxis
* Emergency room visit or hospitalization for severe asthma within 6 months prior to study entry
* HIV-1 infected
* Hepatitis C virus infected
* Hepatitis B surface antigen positive
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive drugs within 30 days prior to study entry. Participants who have used topical or nasal corticosteroids are not excluded.
* Live vaccine within 4 weeks prior to study entry
* Killed vaccine within 2 weeks prior to study entry
* Blood products within 6 months prior to study entry
* Investigational drug or vaccine within 3 months prior to study entry
* Previously received a licensed or experimental yellow fever, tick-borne encephalitis, or dengue vaccine
* Surgical removal of spleen
* History of tick-borne encephalitis
* History of dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis, West Nile virus, Japanese encephalitis virus)
* Other condition that, in the opinion of the investigator, would affect the participant's participation in the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2005-07; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related adverse effects, graded by intensity and severity through active and passive surveillance | Throughout study
Immunogenicity of vaccine against anti-Langat neutralizing antibody | At Days 0, 28, 42, and 180

SECONDARY OUTCOMES:
Recovery of virus from the blood of a vaccinee or seroconversion | Throughout study
Immunogenicity of the LGT(TP21)/DEN4 vaccine against other TBE viruses | Throughout study
Durability of antibody responses to Langat and other TBE viruses | At Day 180

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research, Johns Hopkins School of Public Health; Peter Wright, MD, Principal Investigator — Vanderbilt University School of Medicine
Locations (1):
- Vanderbilt University School of Medicine, Nashville, Tennessee, United States

REFERENCES:
- [Background] Beran J. Immunisation against tick-borne encephalitis by widely used vaccines: short-term history and current recommendations. Clin Microbiol Infect. 2005 May;11(5):424-6. doi: 10.1111/j.1469-0691.2005.01115.x. No abstract available. PMID 15819877
- [Background] Chang GJ, Kuno G, Purdy DE, Davis BS. Recent advancement in flavivirus vaccine development. Expert Rev Vaccines. 2004 Apr;3(2):199-220. doi: 10.1586/14760584.3.2.199. PMID 15056045
- [Background] Lai CJ, Monath TP. Chimeric flaviviruses: novel vaccines against dengue fever, tick-borne encephalitis, and Japanese encephalitis. Adv Virus Res. 2003;61:469-509. doi: 10.1016/s0065-3527(03)61013-4. PMID 14714441
- [Background] Pletnev AG, Bray M, Hanley KA, Speicher J, Elkins R. Tick-borne Langat/mosquito-borne dengue flavivirus chimera, a candidate live attenuated vaccine for protection against disease caused by members of the tick-borne encephalitis virus complex: evaluation in rhesus monkeys and in mosquitoes. J Virol. 2001 Sep;75(17):8259-67. doi: 10.1128/jvi.75.17.8259-8267.2001. PMID 11483771